CLINICAL TRIAL: NCT00130962
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of ALGRX 4975 in Subjects With Painful Intermetatarsal Neuroma
Brief Title: ALGRX 4975 in the Treatment of Patients With Morton's Neuroma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoRx Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4975-2-004-1
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2005-10-03 (Estimated); Status verified 2005-08

CONDITIONS: Neuroma
Keywords: Intermetatarsal neuroma; Morton's neuroma; ALGRX 4975; capsaicin
MeSH Terms: conditions — Neuroma; Morton Neuroma

INTERVENTIONS:
Drug: ALGRX 4975

SUMMARY:
Subjects will have painful primary or post-operative intermetatarsal neuroma. Study drug or placebo will be injected into the space containing the neuroma. Subjects will complete weekly assessments for severity of foot pain, a brief pain inventory, and the amount of pain medication taken. Subjects will be seen for a screening visit, a treatment visit, and two follow-up visits after treatment. The last scheduled visit is one month after treatment. Some subjects may be followed by monthly telephone interviews to assess their level of pain over the six-month period following treatment.

DETAILED DESCRIPTION:
Subjects will have painful primary or post-operative intermetatarsal neuroma. Each subject will be randomly allocated to receive either ALGRX 4975 or placebo in a 1:1 ratio. Study drug or placebo will be injected into the intermetatarsal space containing a painful neuroma. Subjects will complete weekly assessments for the Average Foot Pain Severity, the 7 Interference Items of the BPI, and the number of analgesic units taken. Some subjects may be followed by monthly telephone interviews to assess their level of pain over the six-month period following treatment.

Plasma concentrations will be assessed pre-dose and post dose at 5, 10, 15, 20, 30, and 45 min and at 1, 1.5, 2, 2.5, 3 and 4 hours.

Safety will be assessed at baseline and during the study with adverse events (all visits), vital signs (Visit 2 pre and post-injection and Visit 3 or at early termination), and laboratory assessments (hematology, chemistry, urinalysis) and ECG (Screening and Visit 3 or at early termination). The injection site will be examined and assessed by a 6-point scale for erythema, edema, and hemorrhage before the injection and at 1, 2 and 4 hours after the injection. A pain on injection NRS will be assessed immediately post- injection at 15, 30, and 45 minutes and 1, 2, 3, and 4 hours after study drug administration. A sensory examination of the foot will be performed before the injection and 4 hours after the injection and at the completion of the study. If a subject has injection pain, the foot may be wrapped in ice for up to 20 minutes, analgesic medication may be provided.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged >18 years
* Foot X-ray to rule out alternative pathology, and ultrasound or magnetic resonance imaging (MRI) to confirm the presence of a neuroma within 6 months of study entry
* Evidence of either a primary or post surgical recurrence neuroma
* A score of 4 or greater on the Average Foot Pain Severity Numeric Rating Scale (NRS) during the week prior to randomization
* Failed conservative treatment such as wide shoes, orthotics, arch supports, or oral and/or injected analgesics
* Signed an Informed Consent form approved by the Institutional Review Board
* For female subjects: is surgically sterile, at least 2 years postmenopausal, or using a medically acceptable method (as determined by the Principal Investigator) of birth control; if of child-bearing potential is not pregnant (have a documented negative urine pregnancy test prior to enrollment), is not planning to get pregnant (during the time course of the study), or is not lactating
* Able to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments

Exclusion Criteria:

* History of clearly documented allergic reaction to lidocaine or capsaicin.
* Prior participation in ALGRX 4975 study.
* Presence of any medical condition or instability that, in the judgment of the Investigator, might adversely impact the conduct of the study and the collection of data, including chronic conditions that are likely to alter the rate of healing or are likely to result in safety complications unrelated to the study medication, such as diabetes mellitus or extensive vascular disease
* Treatment of neuroma with a narcotic analgesic
* Other painful foot pathology
* Active cutaneous, or other disease, at the anticipated site of study drug injection
* Laboratory results that are both out of normal range and, in the opinion of the Investigator, clinically significant
* Drug or alcohol abuse within the past 2 years
* Require regular oral steroid medication, except for stable use (6 months or longer on the same scheduled dose) for mild or moderate asthma
* Use of an investigational medication in the 30 days prior to the current study or scheduled to receive such an agent while participating in the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2006-02

PRIMARY OUTCOMES:
Weekly average foot pain severity scores

SECONDARY OUTCOMES:
The sum of weekly average foot pain severity scores
Interference item scores of the Brief Pain Inventory
Weekly number of analgesic units taken

CONTACTS AND LOCATIONS:
Overall Officials: Eric Diamond, D.P.M., Principal Investigator — Crossroads Research, Inc.
Locations (2):
- United States (2):
  - Crossroads Research, Inc., Owings Mills, Maryland
  - Jean Brown Research, Salt Lake City, Utah